CLINICAL TRIAL: NCT07174505
Title: A Prospective, Single-Arm, Multi-Center Study to Assess the Safety, Performance, and Preliminary Efficacy of Mechanical Thrombectomy Using the CONDA Stent Retriever in Subjects With Acute Ischemic Stroke
Brief Title: Evaluation of the CONDA Stent Retriever in Acute Ischemic Stroke
Acronym: ARTEMIS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Anaconda Biomed S.L. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CON2501
Record Dates: First submitted 2025-09-11; First posted 2025-09-16 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Acute Ischemic Stroke; Large Vessel Occlusion
Keywords: Acute Ischemic Stroke (AIS); mechanical thrombectomy; stent retriever
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Masking Description: Independent imaging core will evaluate reperfusion outcomes
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CONDA Device (Experimental): The CONDA device is a stent retriever intended to enable the entrapment and removal of clotted blood in the neurovasculature in subjects experiencing acute ischemic stroke (AIS) secondary to large vessel occlusion (LVO) and treated within 24 hours of symptom onset. All participants in the study will receive Mechanical Thrombectomy using the device following standard of care practice for neurovascular procedures.
  Interventions: Device: Mechanical Thrombectomy using the CONDA Stent Retriever

INTERVENTIONS:
Device: Mechanical Thrombectomy using the CONDA Stent Retriever — Intravenous sedation, local or general anesthesia, and anticoagulation management will be administered following the institution's standard of care to ensure subject safety and comfort. These procedures should be applied to the target population at the discretion of the investigator and in accordance with clinical guidelines. The use of CONDA is no different than that established for other CE marked stent retrievers. The use of supportive devices including, long sheaths, guide catheters with our without balloons, distal access catheters, ANA funnel catheter, microcatheters and microwires, along with the CONDA device, will be guided by operator preference and/or center established practices. Operators are required to use these devices according to their labeling and instructions for use.

SUMMARY:
The goal of this study is to evaluate the safety and performance of the CONDA stent retriever in patients with acute ischemic stroke due to large vessel occlusion, treated within 24 hours of symptom onset.

The main objectives are:

* To determine the rate of device success, defined as the ability of the CONDA retriever to reach the blocked vessel, be deployed and retrieved successfully, and facilitate reperfusion.
* To evaluate safety, measured as the rate of symptomatic intracranial hemorrhage within 24 hours of the procedure.

The use of CONDA in this study follows the same approach as other CE-marked stent retrievers. Supportive devices (such as long sheaths, guide catheters, balloon catheters, distal access catheters, the ANA funnel catheter, microcatheters, and microwires) may be used according to investigator preference and local practice, in line with their labeling and instructions for use.

Participants will:

* Be evaluated using standard clinical and imaging assessments to confirm eligibility.
* Undergo mechanical thrombectomy with the CONDA device, with or without supportive devices as selected by the treating physician.
* Have standard follow-up evaluations to assess treatment safety and effectiveness.

DETAILED DESCRIPTION:
ARTEMIS is a pilot prospective, multi-center, single-arm, open-label, interventional study. Standard of care clinical and imaging stroke assessments will determine subject eligibility. The objective of this study is to assess the performance, safety and preliminary efficacy of mechanical thrombectomy (MT) using the CONDA device in its intended use as a stent retriever to enable the entrapment and removal of clotted blood in the neurovasculature in subjects experiencing acute ischemic stroke (AIS) secondary to large vessel occlusion (LVO) and treated within 24 hours of symptom onset. The ARTEMIS study is designed to demonstrate that the use of CONDA does not adversely impact the safety and effectiveness of a conventional stent retriever MT procedures.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 to 85 years.
2. Informed consent was obtained from subject or acceptable subject surrogate (e.g., next of kin, or legal representative).
3. New focal disabling neurologic deficit consistent with acute cerebral ischemia.
4. Baseline NIHSS obtained prior to procedure ≥ 6 points and ≤ 25 points.
5. Pre-ictal mRS score of 0, 1 or 2.
6. Treatable within 24 hours of stroke symptom onset.
7. If indicated, thrombolytic therapy shall be initiated following recommendations established by the AHA/ASA and/or ESO Guidelines. Subjects eligible for IV thrombolysis should receive it without delay.
8. Extended Thrombolysis in Cerebral Infarction (eTICI) Score 0 - 1, confirmed by angiography or CTA/MRA of the:

   1. Intracranial internal carotid artery (ICA)
   2. Middle cerebral artery - M1 segment
   3. Middle cerebral artery - M2 proximal or dominant segments
9. Imaging criteria:

   * Alberta Stroke Program Early CT Score (ASPECTS) 6 to 10 on baseline CT or DWI-MRI.
   * If automated assessment, core volume of ≤50 cc on CTP/ DWI-MRI.

Exclusion Criteria:

The following exclusion criteria will be assessed pre-operatively:

1. Rapid neurological improvement prior to enrollment suggesting resolution of stroke.
2. Subject was diagnosed with a stroke in the last 6 months.
3. Clinical symptoms suggestive of bilateral stroke or stroke in multiple territories.
4. Clinical presentation suggests subarachnoid hemorrhage.
5. Known hemorrhagic diathesis, coagulation factor deficiency, or oral anticoagulant therapy with antivitamin K, with INR >3.0.
6. Known baseline glucose of <50 mg/dL or >400 mg/dL.
7. Severe, sustained uncontrolled hypertension refractory to treatment (systolic blood pressure >185 mmHg or diastolic blood pressure >110 mmHg).
8. Serious, advanced, or terminal disease with anticipated life expectancy of less than 1 year.
9. Known history of severe sensitivity (more than rash) to contrast medium.
10. Known history of severe sensitivity to nickel, titanium metals or their alloys.
11. Known renal insufficiency with creatinine ≥3 mg/dL or glomerular filtration rate (GFR) <30 mL/min.
12. Subject requires hemodialysis or peritoneal dialysis.
13. Subject is a current user or has a recent history of cocaine and/or heroin use.
14. Known pregnancy and/or lactating female.
15. Subject is participating in a concurrent study involving an investigational drug or device that would impact the primary endpoint of this study.
16. Subject is unlikely to be available for a 90-day follow-up (e.g., no fixed home address, visitor from overseas, etc.)
17. CT or MRI evidence of hemorrhage (the presence of microbleeds is allowed).
18. CT or MRI evidence of significant mass effect with midline shift.
19. CT or MRI evidence of intracranial tumor (except asymptomatic meningioma of ≤ 2cm in diameter).
20. CT or MR evidence of cerebral vasculitis.
21. Suspicion of aortic dissection, presumed septic embolus, or bacterial endocarditis.
22. History of preexisting stent proximal to or at the occlusion site that may preclude safe deployment or recovery of the stent retriever.

    The following exclusion criteria will be assessed intra-operatively:
23. eTICI score improvement to greater than eTICI 1 after initial screening and prior to intervention.
24. Initially treated with a different thrombectomy device during the current study procedure.
25. Vessel tortuosity too difficult to allow endovascular access of the intracranial internal carotid artery (ICA) per investigator judgement. Indicators of vessel tortuosity include but are not limited to the presence of carotid loops and type 3 aortic arches.
26. Evidence of tandem lesions, including complete occlusion, high-grade stenosis or arterial dissection in the extracranial or intracranial internal carotid artery (ICA), requiring treatment or preventing access to thrombus.
27. Underlying intracranial atherosclerotic disease (ICAD) lesions responsible for the target occlusion.
28. Occlusions in multiple vascular territories (e.g., bilateral anterior circulation, or anterior/posterior circulation).
29. Inability to gain arterial access.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2026-10-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Rate of device success | Day 0 Index Procedure
  The rate of device success is defined as the ability of the CONDA retriever to reach the target occluded vessel, be deployed and retrieved successfully, while facilitating reperfusion. Success will be determined if both of the following criteria are met: a) Device Performance, b) Clinical Performance
Incidence of symptomatic intracranial hemorrhage | 24 hours (-8/+12) of the index procedure
  (sICH) defined per SITS-MOST criteria, attributable to the device or procedure, occurring within 24 hours (-8/+12) of the index procedure and assessed by the Imaging Core Lab and Data Monitoring Committee (DMC).

CONTACTS AND LOCATIONS:
Locations (2):
- Semmelweis University Hospital, Budapest, Hungary
- Vall d'Hebron University Hospital, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Undecided